CLINICAL TRIAL: NCT04034563
Title: Post-polypectomy Surveillance Interval In High-risk Subjects After Screening Colonoscopy (PPSHR).
Brief Title: Post-polypectomy Surveillance Interval In High-risk Subjects After Screening Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joseph JY SUNG, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPSHR_PROTOCOL_Ver.1_20170405
Record Dates: First submitted 2019-04-16; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Surveillance Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk of advanced neoplasia at 3-year (Other): Risk of metachronous advanced neoplasia in those patients who done surveillance colonoscopy at 3-years
  Interventions: Procedure: 1) Risk of metachronous advanced neoplasia at 3-year, beyond 3 years surveillance colonoscopy
- Risk of advanced neoplasia beyond 3-year (Other): Risk of metachronous advanced neoplasia in those patients who done surveillance colonoscopy beyond 3-years
  Interventions: Procedure: 1) Risk of metachronous advanced neoplasia at 3-year, beyond 3 years surveillance colonoscopy

INTERVENTIONS:
Procedure: 1) Risk of metachronous advanced neoplasia at 3-year, beyond 3 years surveillance colonoscopy — 3-year group: High-risk subjects who have baseline colonoscopy done in 2014, 2015 and 2016 and will be eligible for 3-year surveillance colonoscopy in 2017-2019.
  Beyond 3 years group: High-risk subjects who had screening colonoscopy prior 3 years, but not received or scheduled for a surveillance colonoscopy- either due to non-adherence or limited access to surveillance colonoscopy will be eligible for surveillance colonoscopy in 2017-2019.
  For the surveillance interval beyond 3 years group, recruitment will be prioritizing to subjects who had the screening colonoscopy at the earliest date. This will in part ensure that subjects in this group will consist those with the longest surveillance interval, leading to an applicable estimation of the risk of metachronous advanced neoplasia beyond 3 years surveillance interval.

SUMMARY:
With many countries initiating population colorectal cancer (CRC) screening, including Hong Kong, more robust guidance for surveillance interval is required to maximize subject's benefit with optimal use of resources. Surveillance interval after removal of advanced adenoma at screening colonoscopy remains unclear. The current recommendation of 3-year is based on data collected before widespread implementation of population screening programs and quality metrics in colonoscopy. These high-risk subjects are those most likely to benefit from surveillance and represent the majority of the demand in surveillance colonoscopies.

DETAILED DESCRIPTION:
The aim of the study is to determine whether the risk of metachronous advanced neoplasia increases if surveillance interval was beyond the current recommendation of 3 years for high-risk subjects with advanced adenoma polyp at screening colonoscopy.

With many countries initiating population colorectal cancer (CRC) screening, including Hong Kong, more robust guidance for surveillance interval is required to maximize subject's benefit with optimal use of resources. Surveillance interval after removal of advanced adenoma at screening colonoscopy remains unclear. The current recommendation of 3-year is based on data collected before widespread implementation of population screening programs and quality metrics in colonoscopy. These high-risk subjects are those most likely to benefit from surveillance and represent the majority of the demand in surveillance colonoscopies.

The investigators hypothesize that the risk of metachronous advanced neoplasia significantly increases if surveillance interval was prolonged beyond 3 years for high-risk subjects. If such is true, our study's findings will provide definitive evidence to existing guidelines and the future Hong Kong population CRC screening programme of setting surveillance interval at 3-year. Conversely, if our study shows that there is no significant increase in risk beyond 3-year surveillance interval, an extended interval of 5-year is justified.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced adenoma at screening colonoscopy
2. ≥3 adenomas at screening colonoscopy
3. Cecal intubation at screening colonoscopy (preferably documented by images/video of the apendiceal orifice and the ileocecal valve; but not required)
4. Complete excision of all polyps at screening colonoscopy findings (after review of endoscopy reports and pathological specimens)
5. Eligible for surveillance in out-patient setting

Exclusion Criteria:

1. Lack of consent
2. Incomplete screening colonoscopy
3. Incomplete endoscopic excision of polyps at screening colonoscopy
4. CRC at screening colonoscopy
5. Polyps requiring Endoscopic Submucosal Dissection at screening colonoscopy
6. Serrated polyps ≥ 10 mm in diameter at any colorectal location or ≥ 5 mm if located proximal to the splenic flexure on screening colonoscopy
7. Genetic cancer syndrome (adenomatous or serrated polyposis syndrome; Lynch or Lynch-like syndrome)
8. Inflammatory bowel disease
9. History of surgical colon resection for any reason
10. Severe co-morbidity with reduced life expectancy (NYHA 3-4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Advanced neoplasia detection rate | Up to 3 months
  Advanced neoplasia detection rate in surveillance colonoscopy among the two groups of patients

SECONDARY OUTCOMES:
CRC detection rate | Up to 3 months
  CRC detection rate in surveillance colonoscopy among the two groups of patients

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Endoscopy Center, Prince of Wales Hospital, Hong Kong
  - S.H. Ho Centre for Digestive Health, Prince of Wales Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No